CLINICAL TRIAL: NCT00464321
Title: A Phase I, Multicentre, Open-label, Dose-escalating Study of Single Doses of GC1008 in Patients With Treatment Resistant Idiopathic Focal Segmental Glomerulosclerosis (FSGS)
Brief Title: Safety Study of GC1008 in Patients With Focal Segmental Glomerulosclerosis (FSGS) of Single Doses of GC1008 in Patients With Treatment Resistant Idiopathic FSGS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC1008FSGS00505
Record Dates: First submitted 2007-04-20; First posted 2007-04-23 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-03

CONDITIONS: Focal Segmental Glomerulosclerosis
MeSH Terms: conditions — Glomerulosclerosis, Focal Segmental | interventions — fresolimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort A (Experimental): Dose Group
  Interventions: Biological: GC1008
- Cohort B (Experimental): Dose Group
  Interventions: Biological: GC1008
- Cohort C (Experimental): Dose Group
  Interventions: Biological: GC1008
- Cohort D (Experimental): Dose Group
  Interventions: Biological: GC1008

INTERVENTIONS:
Biological: GC1008 — 1 mg/kg, IV infusion on Day 0 and monitored over 24 hours. Post infusion for safety up to 112 days.
  Arms: Cohort A
Biological: GC1008 — 2 mg/kg, IV infusion on Day 0 and monitored over 24 hours. Post infusion for safety up to 112 days.
  Arms: Cohort B
Biological: GC1008 — 4 mg/kg, IV infusion on Day 0 and monitored over 24 hours. Post infusion for safety up to 112 days.
  Arms: Cohort C
Biological: GC1008 — 0.3 mg/kg, IV infusion on Day 0 and monitored over 24 hours. Post infusion for safety up to 112 days.
  Arms: Cohort D

SUMMARY:
This study will investigate whether GC1008, an antibody which neutralizes TGF-beta, is safe in treating patients with the disease called focal segmental glomerulosclerosis (FSGS). The highest dose without excessive side effects will be investigated. Tests will determine how long GC1008 is in the body and how it is excreted.

DETAILED DESCRIPTION:
Patients in each cohort will receive a single dose of GC1008 infusion at 1, 2, 4 or 0.3 mg/kg body weight. The higher dose cohort will not start until the first 28 days safety data for the lower dose cohort have been reviewed by the independent Data Monitoring Committee (DMC). Cohort C and D will run concurrently with patients randomised to receive either a 4 or 0.3 mg/kg body weight dose, respectively. After receiving the infusion of GC1008 on Day 0, patients will be monitored for the 24 hours following the infusion. Patients will return periodically over the following 112 days for safety evaluations and clinical outcome assessments. Blood samples will be collected to evaluate the pharmacokinetics of single dose administration of GC1008 as well as for evaluation of markers of clinical efficacy

ELIGIBILITY:
Inclusion Criteria:

* GFR≥25ml/min/1.73m2 calculated by the MDRD equation
* Urinary total protein: creatinine ratios >200mg/mmol derived from the average of 2 first morning voids taken during screening period
* Biopsy confirmed as idiopathic FSGS by a central reviewer
* Treatment resistance. NOTE:Patients to have received minimum 6 week course of steroids or immunosuppressant
* If receiving treatment with an ACEi and/or ARB dose to be stable for a minimum of 4 weeks prior to randomization
* Influenza vaccine (according to season)
* Negative screening per American Cancer Society (ACS) 2003 guidelines, as appropriate to patient demographics and clinical status

Exclusion Criteria:

* Secondary FSGS
* steroid resistant patients who are unable to reduce their steroid dose to <10mg/day of prednisolone or equivalent 4 weeks prior to study dosing day
* Positive serology for serious infections (including but not limited to infection with Hep B or C, HIV)
* Concomitant illnesses:Diabetes Type I; Cardiac or Hepatic disease, HIV; Cancer, precancerous state (eg familial adenomatous polyposis; Any condition requiring treatment with other immunosuppressant drugs within 4 weeks prior to dosing day or during the course of the study
* Pre-existing oral-pharyngeal disease (dental carries and other minor dental disease are acceptable)
* Haemoglobin level of <9.0g/dL prior to dosing
* Treatment with coumadin, anti-vitamin K analogues or low molecular weight heparins. Patients must have stopped treatment a minimum of four weeks prior to receiving study medication.
* Patients requiring ongoing treatment with non-steroidal anti-inflammatory drugs (NSAIDs). Patients must have stopped treatment a minimum of four weeks prior to receiving study medication.
* Patients who have had surgery/fracture within 3 months prior to dosing day
* History of cancer unresolved within 5 years prior to screening or a known precancerous state; or any form of skin cancer either current or past history
* Women who are pregnant, lactating or who plan to become pregnant within 4 months of infusion
* Women of childbearing potential unless taking medically acceptable contraceptive
* Men with female partners of childbearing potential unless they are taking medically acceptable contraceptive precautions
* Use of any investigation drug administered as part of a clinical trial within 4 weeks prior to commencing screening
* Other clinically significant, uncontrolled medical condition that in the investigator's opinion may interfere with the assessment or follow-up
* Active ethanol or drug abuse, excluding tobacco use
* Electrocardiogram (ECG) abnormalities considered to be clinically significant at screening
* Unable to comply with the requirements of the study
* Active thrombophlebitis, thromboembolism, hypercoagulability states, bleeding, or use of anticoagulation therapy (including anti-platelet agents). Patients with a history of deep venous thrombosis may participate if successfully treated, completely resolved, and no treatment has been given for >4 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-05; Primary Completion 2010-01 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
To determine Safety and tolerability of single dose infusions of GC1008 in patients with treatment resistant idiopathic FSGS and nephrotic range proteinuria | up to 2 years
Pharmacokinetics of GC1008 following a single dose infusion | up to 2 years

SECONDARY OUTCOMES:
To investigate Effect of single dose infusions of GC1008 on biomarkers of clinical efficacy. | up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (9):
- United States (4):
  - San Francisco, California
  - Rochester, Minnesota
  - New Hyde Park, New York
  - Chapel Hill, North Carolina
- Germany (3):
  - Berlin
  - Düsseldorf
  - Solingen
- Bergamo, Italy
- Cambridge, United Kingdom